CLINICAL TRIAL: NCT05781711
Title: Clinical Study to Evaluate the Possible Efficacy of Metformin in Patients With Parkinson's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Manal Ali Mahrous Hamouda Faculty of Pharmacy, Menufia University (Unknown)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2023
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Control group ( Levo-dopa group, n =30 ) who will receive levodopa/carbidopa (50/250 mg) three times daily for 3 months
  Interventions: Drug: levodopa-carbidopa
- Metformin group (Active Comparator): Patients will receive levodopa/carbidopa (50/250 mg) three times daily plus metformin 500 mg two times daily for 3 months
  Interventions: Drug: levodopa-carbidopa; Drug: Metformin

INTERVENTIONS:
Drug: levodopa-carbidopa — levodopa-carbidopa is the standard therapy used in Parkinson's disease
Drug: Metformin — Metformin, a biguanide family member commonly used in treatment for type 2 diabetes, appears to increase liver and peripheral tissue sensitivity to insulin as well as reduce hepatic glucose production
  Arms: Metformin group

SUMMARY:
Parkinson's disease (PD) is one of the most common neurodegenerative diseases characterized by the progressive loss of dopaminergic (DA) neurons in the substantia nigra compacta (SNc) and aggregation of Lewy bodies in neurons. Although aging, oxidative damage and neuroinflammation have been recognized to play crucial roles in the pathogenesis of PD, the precise etiology remains obscure. Emerging evidence suggests PD is a systemic metabolic disease, and metabolic abnormality correlates with functional alternations in PD

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Both males and females will be included Negative pregnancy test and effective contraception. Diagnosed Parkinson's disease patient taking Levodopa

Exclusion Criteria:

Secondary causes of Parkinsonism Diabetic patients Patients taking anti-inflammatory drugs Atypical parkinsonian syndromes Prior stereotaxic surgery for Parkinson's disease Pregnancy and lactation Suffering from active malignancy Addiction to alcohol and/or drugs Known allergy to the studied medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
• The primary endpoint is the change in The Unified Parkinson's Disease Rating Scale (UPDRS) | 3 months
  • The primary endpoint is the change in the Unified Parkinson's Disease Rating Scale (UPDRS

SECONDARY OUTCOMES:
The secondary endpoint is estimated by changes in serum biomarkers. | 3 months
  The secondary endpoint is estimated by changes in serum biomarkers such as brain derived neurotropic factor

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Menoufia University, Tanta, Shebeen El-Kom, Egypt

REFERENCES:
- [Derived] AlRasheed HA, Bahaa MM, Elmasry TA, Elberri EI, Kotkata FA, El Sabaa RM, Elmorsi YM, Kamel MM, Negm WA, Hamouda AO, Aldossary KM, Salahuddin MM, Yasser M, Eldesouqui M, Hamouda MA, Eltantawy N, Elawady ME, Abdallah MS. Randomized, double-blind, placebo-controlled pilot study of metformin as an adjunctive therapy in Parkinson's disease. Front Pharmacol. 2025 May 2;16:1497261. doi: 10.3389/fphar.2025.1497261. eCollection 2025. PMID 40385486